CLINICAL TRIAL: NCT00378625
Title: Randomised, Double Blind Clinical Trial of the Efficacy, Effect on Gametocytes and Tolerability of Amodiaquine Vs Amodiaquine Plus Artesunate in the Treatment of Uncomplicated P. Falciparum Malaria in Quibdo, Colombia
Brief Title: Efficacy, Effect on Gametocytes and Tolerability of the Addition of Artesunate to Amodiaquine in Colombia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centro Internacional de Entrenamiento e Investigaciones Médicas (Other)
Collaborators: World Health Organization (Other); Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: A00096/990954; 2229-04-10380
Record Dates: First submitted 2006-09-18; First posted 2006-09-20 (Estimated); Last update posted 2006-09-20 (Estimated); Status verified 2006-09

CONDITIONS: Malaria,Falciparum; Malaria; Antimalarials
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Artesunate

INTERVENTIONS:
Drug: Artesunate

SUMMARY:
The primary goal of this study is to quantify the benefit of adding artesunate to amodiaquine in treating patients with uncomplicated P. falciparum malaria, in a low transmission area in Colombia. The benefit will be assessed in terms of:

* Efficacy
* Tolerability
* Time of fever clearance
* Time of parasite clearance
* Proportion of gametocyte carriers

ELIGIBILITY:
Inclusion Criteria:

1. pure P. falciparum infection
2. parasitaemia >500 and <50,000 asexual parasites/μL (subsequently the lower limit was modified to >250 asexual parasites/μL)
3. age between 1 and 65 years old
4. availability to return for follow-up

Exclusion Criteria:

1. Pregnancy
2. history of allergy to the study drugs
3. history of taken complete treatment with an antimalarial drug in the previous 72 hours or sulphas, clindamycin or tetracycline in the previous week
4. have a medical history of untreated hypertension or chronic heart, kidney or liver disease
5. present any danger signs of severe malaria.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360
Dates: Start 2000-04; Study Completion 2006-03

PRIMARY OUTCOMES:
treatment failures
adverse events
gametocyte carriage

CONTACTS AND LOCATIONS:
Overall Officials: Lyda Osorio, MD PhD, Principal Investigator — Centro Internacional de Entrenamiento e Investigaciones Médicas
Locations (1):
- Hospital Ismael Roldan and Centro de Salud San Vicente, Quibdó, Departamento del Chocó, Colombia